CLINICAL TRIAL: NCT04657822
Title: An Open-label, Multi-center, Phase IV, Rollover Study for Patients With Sickle Cell Disease Who Have Completed a Prior Novartis-Sponsored Crizanlizumab Study
Brief Title: Rollover Study for Patients With Sickle Cell Disease Who Have Completed a Prior Novartis-Sponsored Crizanlizumab Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSEG101A2401B; 2020-004225-22 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
Keywords: SCD; Vaso-occlusive Crisis; crizanlizumab; SEG101; Sickle cell disease; Sickle cell disorder; VOC; P-selectin; Sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — crizanlizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crizanlizumab (Experimental): All participants will receive crizanlizumab (SEG101) at the same dose/schedule as in the parent study.
  Interventions: Drug: Crizanlizumab

INTERVENTIONS:
Drug: Crizanlizumab — Concentrate for solution for infusion for Intravenous use
  Other Names: SEG101

SUMMARY:
This is a multi-center multi-national rollover study to allow continued access to crizanlizumab for patients with sickle cell disease (SCD) who are on crizanlizumab treatment in a Novartis-sponsored study (parent study) and are benefiting from the treatment as judged by the investigator.

DETAILED DESCRIPTION:
There will be no screening period for this study as patients will transfer directly from parent studies. After providing informed consent, all eligible participants should start Crizanlizumab treatment at the earliest convenience following the treatment schedule of 28 days of the last dose in the parent study. Crizanlizumab will be administered at the same dose/schedule as in the parent study.

Study participants will have a safety follow up visit conducted 105 days after last administration of study treatment. The safety follow up at 105 days is not applicable for those participants who continue to receive Crizanlizumab after end of treatment visit either commercially or through PSDS.

The study is expected to remain open for 10 years from the first Patient's first visit (FPFV) in this clinical study or until study treatment becomes commercially available and is reimbursed in the respective indication or until such time that all enrolled patients no longer need treatment with Crizanlizumab, or a PSDS treatment plan is allowed and approved as per local laws and regulations, whichever comes first

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent, according to local guidelines, signed by the adult patients. In the population under 18 years, it will be signed by the patient and/or by the parents or legal guardian prior to enrolling in the rollover study and receiving study medication
2. SCD patient currently enrolled in a Novartis-sponsored study receiving crizanlizumab and has fulfilled all the requirements in the parent study. Patient is currently benefiting from the treatment with crizanlizumab as determined by the investigator and has completed the treatment schedule as planned in the parent study
3. Patient has demonstrated compliance to the planned visit schedule in the parent study, and in the opinion of the investigator has shown willingness and ability to comply with future visit schedules

Exclusion Criteria:

1. Patient had permanently discontinued from crizanlizumab study treatment in the parent study before the parent study completion
2. Ongoing/unresolved treatment-related Grade 3 or higher AEs, and/or any ongoing AE requiring dose interruption. Patients meeting all other eligibility criteria may be enrolled once toxicities have resolved unless those toxicities were grade 4
3. Concurrent participation in any other investigational clinical trial other than the parent study or plan to participate in any other investigational clinical trial
4. Pregnant or nursing women
5. Women of childbearing potential who are unwilling to be on highly effective contraceptives during dosing and until 15 weeks after stopping treatment with crizanlizumab
6. SCD patients who do not meet parent study protocol criteria to continue with crizanlizumab

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2031-06-10 (Estimated); Study Completion 2031-06-10 (Estimated)

PRIMARY OUTCOMES:
Not Applicable as this protocol is to provide an option for continued access to crizanlizumab for patients with Sickle Cell Disease who have completed a prior Novartis-sponsored Crizanlizumab study | Not Applicable - Study Completion
  Protocol to provide an option for continued access to crizanlizumab for patients with Sickle Cell Disease who have completed a prior Novartis-sponsored Crizanlizumab study, benefited from the treatment and do not have access to reimbursed, commercially available crizanlizumab.

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | from day of first dose of study medication to 105 days after last dose of study medication
  The number of participants with Frequency, severity and causality of treatment emergent adverse events will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (6):
  - University Of Alabama, Birmingham, Alabama
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Augusta University Georgia, Augusta, Georgia
  - East Carolina University, Greenville, North Carolina
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Childrens Medical Center, Fort Worth, Texas
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Liège
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Colombia (2):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Montería
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Heidelberg, Germany
- Italy (2):
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Orbassano, TO
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Tripoli
- Novartis Investigative Site, Khoudh, Oman
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Hatay, Antakya
  - Novartis Investigative Site, Adana, Saricam
  - Novartis Investigative Site, Adana, Yuregir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com